CLINICAL TRIAL: NCT06527196
Title: TEAMS R34 #3: Developing and Testing a Team-Based Implementation Strategy for Depression Screening in a Pediatric Health Care System
Brief Title: TEAMS R34 #3: Team-Based Implementation Strategy for Pediatric Depression Screening
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Nicole Stadnick, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 810627; P50MH126231 (NIH)
Record Dates: First submitted 2024-07-19; First posted 2024-07-30 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Depression; Children
Keywords: Depression Screening; Team Charter; Team Effectiveness
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Condition (Active Comparator): In the comparison condition, staff will continue to use multiple discrete strategies already implemented as apart of the depression screening pathway. These existing strategies include:
  1. Training in the depression screening tool (Patient Health Questionnaire)
  2. Orientation to the clinical pathway (i.e., screening conducted at every urgent care or emergency department visit and every 30 days for all other medical visits)
  3. Expectations for handoff to the next step in the care cascade
  Interventions: Behavioral: Standard Condition
- Team-Enhanced Condition (Experimental): The team-enhanced condition will include:
  1. Two initial 1-hour didactic sessions to develop the team charter.
  2. Biweekly check-ins (15-30 minutes) where the research team will review ongoing use of the team charter with participants and explore any necessary revisions.
  Interventions: Behavioral: Team-Enhanced Condition

INTERVENTIONS:
Behavioral: Team-Enhanced Condition — Participants in the experimental arm (team-enhanced condition) will be asked to participate in the creation and use of a team charter. This will occur over a period of six months.
  Arms: Team-Enhanced Condition
Behavioral: Standard Condition — Providers in the standard condition will be asked to continue practices and response to depression screening as currently implemented by the hospital system.
  Arms: Standard Condition

SUMMARY:
Pediatric depression is a global concern that has fueled efforts for enhanced detection and treatment engagement. While many health systems have implemented components of depression screening protocols, there is limited evidence of effective follow-up for pediatric depression. Key barriers to prompt service linkage include a shared understanding of individual and team member roles and coordination between clinicians and staff across service areas. This project aims to refine and test a team-based implementation strategy, a team charter, improve implementation of an existing pediatric depression screening protocol in a large pediatric healthcare system. The implementation strategy will target team mechanisms at the organizational-level and provider-level. The team charter is hypothesized to lead to improved, efficient, and effective decision-making to increase the frequency of depression screening and timely service linkage. Findings are expected to yield better understanding of how to optimize team activities and patterns in the pediatric depression screening to treatment cascade. This should also culminate in improved patient engagement and outcomes, which are critical to address the youth mental health crisis.

DETAILED DESCRIPTION:
Aim 1: Use mixed methods to refine a team-based implementation strategy to improve implementation of an existing health system universal depression screening protocol (clinical intervention)

Aim 2: Use a two-arm hybrid type 3 implementation-effectiveness pilot trial to assess the initial effectiveness of the team-based implementation strategy on the depression screening protocol.

Aim 3: Use mixed methods to assess team/organizational (intra-organizational alignment, implementation climate) and team member/provider (communication, coordination, psychological safety, shared cognitions) mechanisms of the team-based implementation strategy and a novel application of natural language processing methods.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for all groups of participants are intentionally broad to ensure valid analyses:

1. Employed as medical staff and/or a medical or health provider at Rady Children's Hospital San Diego.
2. Experience providing or supporting care to children and adolescents with mental health care needs.

Exclusion Criteria:

Any individual that does not meet the inclusion criteria will be excluded from study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability, Feasibility, and Appropriateness of Intervention Measure | 6 months
  This 9-item instrument will be administered to participants following completion of the study intervention. The measure was designed to assess the degree to which the intervention is well-received (acceptability), relevant in the given setting (appropriate), and possible and workable (feasibility). The items on the measure (9 total) are each rated on a scale from 1 (completely disagree) to 5 (completely agree). Following completion, individual subscales (3 total) can be obtained by averaging participants' responses for each of the three components (acceptability, appropriateness, and feasibility).
Referral Processing Time | 6 months
  Referral processing, will be based on the time (in hours) from screening to referral based on electronic health record (EHR) timestamps. This will be used to help assess workflow efficiency.
Provider Response Based on Patient Health Questionnaire (PHQ-9) Score | Baseline, 3 months, 6 months
  This measure will be obtained by using the electronic health record (EHR) to determine whether or not providers responded to a patient with an elevated score (10+) on the Patient Health Questionnaire (PHQ-9). This will help researchers assess clinical outcomes of the study intervention (team communication training).
  Context: The Patient Health Questionnaire asks respondents to answer 9 questions that assess mental health status over the patient's last two weeks. Patients answer each question on a scale ranging from 0 (not at all) up to 3 (nearly every day). Scores are calculated by adding individual values together to produce a cumulative score (can range from 0 to 27). A higher score indicates a higher risk for depression symptomology. For the pediatric health system in this study, a score above 10 warrants referral to a behavioral health professional, as well as educational materials and other service referrals.
Mental Health Service Linkage (Caregiver Report of Successful Mental Health Service Linkage) | 3 months, 6 months
  Successful mental health service linkage will be assessed by obtaining caregivers' reports of linkage to any mental health service (internal and external of study's chosen pediatric healthy system) following an elevated depression score on the PHQ-9 (10+).
  Context: The Patient Health Questionnaire asks respondents to answer 9 questions that assess mental health status over the patient's last two weeks. Patients answer each question on a scale ranging from 0 (not at all) up to 3 (nearly every day). Scores are calculated by adding individual values together to produce a cumulative score (can range from 0 to 27). A higher score indicates a higher risk for depression symptomology. For the pediatric health system in this study, a score above 10 warrants referral to a behavioral health professional, as well as educational materials and other service referrals.
Referral Quality (Provider Report of Successful Mental Health Service Referrals) | 6 months
  Referral quality is a measure based on providers' reports of whether referral to the a behavioral health service occurred or not. This will be used to assess workflow efficiency.
Time to Mental Health Service Linkage | Baseline, 3 months, 6 months
  This measure captures time (days) to service linkage for patients that need referrals based on the Patient Health Questionnaire (PHQ-9) score. This data will be obtained from the electronic health record (EHR). This will help researchers assess clinical outcomes of the study intervention (team communication training).
  Context: The Patient Health Questionnaire asks respondents to answer 9 questions that assess mental health status over the patient's last two weeks. Patients answer each question on a scale ranging from 0 (not at all) up to 3 (nearly every day). Scores are calculated by adding individual values together to produce a cumulative score (can range from 0 to 27). A higher score indicates a higher risk for depression symptomology. For the pediatric health system in this study, a score above 10 warrants referral to a behavioral health professional, as well as educational materials and other service referrals.

SECONDARY OUTCOMES:
Implementation Climate Measure | Baseline, 3 months, 6 months
  Implementation climate will be measured with the Implementation Climate Measure. Implementation climate refers to the belief amongst users of an innovation within an organization that utilizing said innovation is rewarded, supported and expected. This instrument consists of 6 items that assess implementation with two questions per climate dimension (expected, supported, and rewarded). The instrument is based on a Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree). Scores are averaged across multiple items to give an overall score or subscale score for implementation climate. Generally, a higher score indicates a more positive perception of implementation climate in an organization. This instrument will be administered to participants through study completion.
Collaboration and Satisfaction About Care Decisions (CSACD) | Baseline, 3 months, 6 months
  The CSACD instrument (6 items total) will be used to assess communication and coordination. For each question, participants respond based on a 7-point likert-type scale where 1= strongly disagree and 7 = strongly agree. 2 individual subscales (3 questions each) can be obtained by averaging responses for the items related to collaboration and the items related to satisfaction.
Card Sorting Activity | Baseline, 3 months, 6 months
  Card sorting is a research assessment to elicit individual mental models about a participant's understanding of a situation, event, or process. Within team contexts, card sorting can be used to interrogate the extent to which team members have aligned thinking about key elements of a situation, event or process, i.e., team mental models.
  In open card sorts participants are given a set of main concepts and told to sort them into different categories. Each makes a specific label for each category. In closed card sorts, participants are also given a set of key concepts, but participants are instead given pre-existing categories to sort concepts into. Each participant from the Aim 2 trial will complete the card-sorting task following team charter development to assess team mental models of member roles, responsibilities, and goals across depression care cascade team members.
Edmonson's Psychological Safety (Interpersonal Risk Taking) Climate Measure | Baseline, 3 months, 6 months
  Psychological safety, which refers to an individual's understanding that the workplace, (specifically the policies/procedures) cultivates a safe arena for interpersonal risk taking, will be measured using Edmonson's Psychological Safety Climate Measure. Participants respond to 7 items total with answer choices from 0 (doesn't apply at all) up to 4 (entirely applies). Scale scores are then determined by averaging responses to each item. Generally, a higher score indicates a stronger perception of psychological safety within the team.
Family Demographics Questionnaire | Baseline, 3 months, 6 months
  Child demographics will be obtained using a Family Demographics Questionnaire and the electronic health record (EHR).

CONTACTS AND LOCATIONS:
Overall Officials: Nicole A Stadnick, PhD, MPH, Principal Investigator — UCSD Associate Professor
Locations (1):
- UC San Diego: IN STEP Children's Mental Health Research Center, San Diego, California, United States

REFERENCES:
- [Derived] Stadnick NA, Aarons GA, Edwards HN, Bryl AW, Kuelbs CL, Helm JL, Brookman-Frazee L. Cluster randomized trial of a team communication training implementation strategy for depression screening in a pediatric healthcare system: a study protocol. Implement Sci Commun. 2024 Oct 18;5(1):117. doi: 10.1186/s43058-024-00641-5. PMID 39425229